CLINICAL TRIAL: NCT03327961
Title: Scaffold Implantation in Emilia-Romagna Plus Multi Absorbable Gears Intra Coronary
Brief Title: Scaffold in Emilia Romagna and in the MAGIC Network
Acronym: SHERPA-MAGIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, University Hospital of Ferrara
Other Study IDs: 170899
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- scaffold: Patients receiving during PCI the implantation of at least one scaffold
  Interventions: Device: scaffold

INTERVENTIONS:
Device: scaffold — implantation of scaffold (eg Magmaris, Desolve, Others)

SUMMARY:
The prospective study will investigate the clinical performance and long-term safety of scaffold implantation in a real world regional setting. The protocol includes two different networks. The first network includes all cath-labs in the Emilia-Romagna region (SHERPA). The second includes the centers partecipating into the MAGIC retrospective study. Both networks joined into the prospective SHERPA-MAGIC project. Investigators from both networks agreed in indications and strategy implanatation described by the protocol. In each center, after IRB approval, the patients will be enrolled according to established criteria.

DETAILED DESCRIPTION:
Coronary stents are the default devices for the treatment of coronary artery disease in percutaneous coronary intervention (PCI) according to existing guidelines. However, thrombosis and restenosis are still the main limitations of current permanent metallic stents. In contrast to Bare Metal Stents (BMSs), Drug Eluting Stents (DESs) have a reduced restenosis rate due to the presence of antiproliferative agents in the coating layer of the stent surface and reduced rate of repeat revascularisation. However, late and very late stent thrombosis remains the limitation of DES in spite of prolonged dual antiplatelet therapy. Bioabsorbable scaffolds have been introduced to overcome limitations of permanent metallic stents.

The aim of this observational prospective study is to investigate the clinical performance and long-term safety of scaffold in a real world regional setting.

The investigators agreed in the following preferential/optimal indications:

* complete revascularization in patients with age <65 years
* revascularization of long lesions (>24 mm), especially located in left anterior descending
* spontaneous coronary dissection

The investigators agreed in the following strategy implantation:

* mandatory predilatation
* sizing 1:1
* to avoid vessel with reference vessel diameter <2.8 mm and >3.8 mm
* to avoid vessel with severe calcifications
* mandatory postdilation with non compliant balloon ≥0.5 the scaffold diameter

The study organization is based on:

DATA SAFETY MONITORING BOARD (DSMB) All adverse events will be reported to the DSMB and reviewed on an on-going basis throughout the subject enrolment and follow-up period to ensure the safety of subjects enrolled in this study. The DSMB may request additional information as needed.

CORE LABORATORY ANALYSIS All coronary artery angiographies and percutaneous coronary interventions will be reviewed by an indipendent core-lab. The core-lab will perform quantitative coronary analysis and assessment of the agreement between implantation technique in each case and established criteria

ELIGIBILITY:
Inclusion Criteria:

* subjects >18 years
* sign of the patients informed consent
* implanation of at least one scaffold

Exclusion Criteria:

* inability to garantuee at least one year follow-up
* inabiliuty to garantuee at least one year compliance to dual antiplatelet regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic coronary artery disease needing the treatment of de novo native coronary artery lesions.
Sampling Method: Non-Probability Sample
Enrollment: 1111 (Estimated)
Dates: Start 2017-12-02 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Device Oriented Cardiac Events | 1 year
  cumulative occurence of cardiovascular death, target vessel myocardial infarction and target vessel revascularization. Target is defined the vessel treated with scaffold

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (17):
  - AO San Giovanni di Dio, Agrigento, Agrigento
  - Ospedale Caravaggio-Treviglio, Treviglio, Bergamo
  - Azienda Ospedaliera Universitaria di Bologna, Bologna, Bologna
  - U.O. Cardiologia, Ospedale Maggiore, Bologna, Bologna
  - Ospedale SS Annunziata, Savigliano, Cuneo
  - University Hospital of Ferrara, Cona, Ferrara
  - U.O. Cardiologia, Ospedale Morgagni Pierantoni, Forlì, Forlì-Cesena
  - U.O. Cardiologia, Azienda Ospedaliera Universitaria di Modena, Policlinico, Modena, Modena
  - U.O. Cardiologia, Ospedale di Baggiovara, Modena, Modena
  - U.O. di Cardiologia, Azienda Ospedaliero-Universitaria di Parma, Parma, Parma
  - Ospedale Guglielmo da Saliceto, Piacenza, Piacenza
  - Maria Cecilia Hospital - GVM Care & Research, Cotignola, Ravenna
  - U.O. di Cardiologia, Ospedale Santa Maria delle Croci, Ravenna, Ravenna
  - U.O. di Cardiologia, Ospedale degli Infermi, Rimini, Rimini
  - AOU San Luigi Gonzaga, Orbassano, Torino
  - Ospedale di Rivoli, Rivoli, Torino
  - Ospedale di Sanremo, Sanremo

IPD SHARING:
Plan to Share IPD: Undecided